CLINICAL TRIAL: NCT00006390
Title: Phase II Study of Campath-1H (NSC #950010) and Peripheral Blood Stem Cell Transplant for Patients With Chronic Lymphocytic Leukemia
Brief Title: Alemtuzumab Plus Peripheral Stem Cell Transplantation in Treating Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068272; ECOG-8998
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Leukemia
Keywords: stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; Filgrastim; Cyclophosphamide; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: alemtuzumab
Biological: filgrastim
Drug: cyclophosphamide
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies such as alemtuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy. Combining monoclonal antibody therapy, chemotherapy, radiation therapy, and peripheral stem cell transplantation may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of alemtuzumab plus peripheral stem cell transplantation in treating patients who have chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the ability of in vivo purging with alemtuzumab (monoclonal antibody CD52; Campath-1H) to produce a stem cell graft without detectable leukemia cells in patients with chronic lymphocytic leukemia.
* Determine the ability to successfully mobilize stem cells after in vivo purging with monoclonal antibody CD52 in these patients.
* Determine the toxicity of this treatment regimen in these patients.
* Determine the response to this treatment regimen in these patients at 6 months after peripheral blood stem cell transplantation.

OUTLINE: This is a multicenter study.

Patients receive induction therapy comprising alemtuzumab (monoclonal antibody CD52; Campath-1H) IV over 2 hours three times a week for 4 weeks.

Beginning no more than 2 weeks after induction therapy, patients receive mobilization chemotherapy comprising cyclophosphamide IV over 1-2 hours on day 1 and filgrastim (G-CSF) subcutaneously (SC) starting on day 2 and continuing until the last day of apheresis. Patients undergo peripheral blood stem cell apheresis on days 10-14.

Beginning 2-4 weeks after apheresis, patients receive a preparative regimen comprising cyclophosphamide IV over 2 hours on days -5 and -4 and fractionated total body irradiation twice a day over 6-10 hours on days -3 to -1. Patients undergo peripheral blood stem cell transplantation on day 0. Patients receive G-CSF SC beginning on day 1 and continuing until blood counts recover.

Patients are followed at 60 days, 1 year, and then annually thereafter until disease progression.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia (CLL) that meets the following criteria at any point prior to study entry:

  * Peripheral blood absolute blood count greater than 5,000/mm^3
  * Lymphocytosis must comprise small to moderate size lymphocytes with no more than 55% prolymphocytes, atypical lymphocytes, or lymphoblasts morphologically
  * Phenotypically characterized B-cell CLL
  * Splenomegaly, hepatomegaly, or lymphadenopathy not required for CLL diagnosis
* Must have bone marrow biopsy within 4 weeks of study entry showing cellularity of at least 25% of intratrabecular space and lymphocytes accounting for no more than 30% of nucleated cells

PATIENT CHARACTERISTICS:

Age:

* 18 to 65

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics
* Absolute neutrophil count at least 1,000/mm^3
* Hemoglobin at least 11 g/dL
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2 mg/dL (unless secondary to tumor)
* AST or ALT less than 3 times upper limit of normal
* Hepatitis B surface antigen negative
* Hepatitis C RNA negative

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* Left ventricular ejection fraction at least 45% by echocardiogram or MUGA

Pulmonary:

* DLCO, FEV_1, and FVC greater than 50% of predicted

Other:

* No active infection requiring oral or IV antibiotics
* No other prior malignancy within the past two years except basal cell skin cancer or carcinoma in situ of the cervix
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior monoclonal antibody CD52 allowed if at least partial remission was achieved with last treatment

Chemotherapy:

* No more than 2 prior chemotherapy regimens
* At least 3 weeks since prior chemotherapy
* No more than 8 courses of prior fludarabine therapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07-05 (Actual); Primary Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian W. Flinn, MD, PhD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (14):
- United States (14):
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Cancer Center at Tufts - New England Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin